CLINICAL TRIAL: NCT00511069
Title: A Phase II Study of Velcade (Bortezomib - PS341) in the Treatment of Patients Over 18 Years With Ph+ Leukemia
Brief Title: Velcade (Bortezomib - PS341) in the Treatment of Patients Over 18 Years With Ph+ Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Bologna (Other)
Responsible Party: Giovanni Martinelli, Dipartimento di Ematologia "seragnoli"- Policlinico Sant'Orsola Bologna
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CML/033-26866138-CAN; EUDRACT 2004-002977-22
Record Dates: First submitted 2007-08-02; First posted 2007-08-03 (Estimated); Last update posted 2008-11-24 (Estimated); Status verified 2008-11

CONDITIONS: Leukemia
Keywords: Bortezomib; CML033
MeSH Terms: conditions — Leukemia | interventions — Bortezomib

INTERVENTIONS:
Drug: Bortezomib

SUMMARY:
Ph+ leukemias (i.e.Chronic Myelogenous Leukemia (CML) and (Ph+) Acute Lymphoblastic Leukemia are malignant clonal disorder of the hemopoietic stem cell due to reciprocal translocation of genetic material between chromosome 9 and 22 giving rise to the translocation t(9;22) (q2.2; q2.1). The translocation causes the formation of a new hybrid gene (bcr-abl) that codes for a 185 kb or 210 kb cytoplasmic protein (P185 and P210 respectively) that by autophosphorylation activates a number of signaling pathways involved in cell proliferation, maturation, apoptosis and adhesion, leading to the malignant cell transformation1-3. The course of the disease goes on through a chronic phase (CP), usually lasting some years, that is characterized by a massive myeloid hyperplasia with hyperleukocytosis and splenomegaly. The CP is almost always followed by an accelerated or blastic phase (ABP) where the leukemic process acquires the characteristics of acute leukemia. The ABP usually lasts some months and terminates with the death of the patient3.

The frequency of CML in western countries ranges between 10 and 15 per million persons (age - standardized). It is rare in children. The median age is 55 years.

Current treatment of CML includes conventional chemotherapy, allogeneic bone marrow transplantation (allo BMT), alpha-interferon (alpha-IFN)and imatinib.

ELIGIBILITY:
Inclusion Criteria for chronic phase patients :

1. Age >/=18 years
2. Ph positive
3. Absence of a CHR after 3 months on imatinib
4. Loss of a previously obtained CHR on imatinib alone
5. Absence of a CCgR within 12 months on imatinib alone
6. Loss of a previously obtained CCgR on imatinib alone
7. Written informed consent

Exclusion Criteria for chronic phase patients :

1. Age <18
2. Performance status (ECOG/WHO) > 2 (see Appendix 2)
3. Inability to provide written informed consent
4. Pregnancy
5. Accelerated or blastic phase
6. Formal refusal of any recommendation of a safe contraception
7. Alcohol or drug addiction
8. Altered hepatic or renal function as defined by AST/ALT or bilirubin > 3 times upper normal limits (UNL)
9. Serum creatinine > 265 umol/l or >3.0 mg/dl
10. Any other disease or condition that by the advise of the responsible physician would make the treatment dangerous for the patient or would make the patient ineligible for the study, including physical, psychiatric, social and behavioural problems.

Inclusion criteria for accelerated and blastic phase or acute lymphoblastic leukemia Ph+ patients:

1. Age >/=18 years
2. Ph positive
3. Loss of a previous hematological response to imatinib alone, with further progression to ABP (see section 14 for definitions)
4. Performance status (ECOG/WHO)
5. Written informed consent

Exclusion criteria for accelerated and blastic phase or acute lymphoblastic leukemia Ph+ patients:

1. Age <18
2. Performance status (ECOG/WHO) > 2 (see Appendix 2)
3. Inability to provide written informed consent
4. Pregnancy
5. Chronic Phase disease
6. Formal refusal of any recommendation of a safe contraception
7. Alcohol or drug addiction
8. Altered hepatic or renal function as defined by AST/ALT or bilirubin > 3 times upper normal limits (UNL)
9. Serum creatinine > 265 umol/l or >3.0 mg/dl
10. Any other disease or condition that by the advise of the responsible physician would make the treatment dangerous for the patient or would make the patient ineligible for the study, including physical, psychiatric, social and behavioural problems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2006-07; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Martinelli, MD, Principal Investigator — Istituto di Ematologia "L e A Seragnoli" Policlinico S.Orsola-Malpighi di Bologna
Locations (1):
- Policlinico "S.Orsola-Malpighi"-Istituto di Ematologia "L e A Seragnoli", Bologna, Italy